CLINICAL TRIAL: NCT05393219
Title: Effects of Preventive Physiological and Psychological Interventions on Performances During Objective Structured Clinical Examination (OSCE) for Medical Students: Cardiac Biofeedback, Mindfulness, or Inner Resources Mobilization
Brief Title: Cardiac Biofeedback, Mindfulness, and Inner Resources Mobilization Interventions on Performances of Medical Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Claude Bernard University (Other)
Responsible Party: Principal Investigator, Lilot Marc, Director, Claude Bernard University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Performance and OSCE
Record Dates: First submitted 2022-05-15; First posted 2022-05-26 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Stress, Psychological; Stress; Stress, Physiological; Exam Stress; Performance; Mindfulness; Communication; Medical Education
MeSH Terms: conditions — Stress, Psychological; Communication | interventions — Mindfulness; Health Resources

STUDY DESIGN:
Intervention Model Description: 4 parallels groups
Who Masked: Investigator, Outcomes Assessor
Masking Description: Performance is evaluated by assessors who are blind to the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cardiac Biofeedback (Experimental): Relaxing breathing exercise coupled with cardiac biofeedback
  Interventions: Other: Cardiac biofeedback
- Mindfulness (Experimental): Mindfulness guided through a video tape
  Interventions: Other: Mindfulness
- Inner resource mobilization (Experimental): Resources and inner strength mobilization guided through a video tape
  Interventions: Other: Resources mobilization
- Control (Sham Comparator): Standardized video tape
  Interventions: Other: Control

INTERVENTIONS:
Other: Cardiac biofeedback — 6 minutes of relaxing breathing exercise coupled with heart rate variability biofeedback guided on emWave Pro software on a computer just before entering the examination circuit
  Other Names: Relaxing breathing exercise coupled with cardiac biofeedback
  Arms: Cardiac Biofeedback
Other: Mindfulness — 6 minutes of a guided video tape made for the study that inspires mindfulness like meditation associated just before entering the examination circuit.
  Other Names: Mindfulness meditation
  Arms: Mindfulness
Other: Resources mobilization — 6 minutes of a guided video tape that purpose to mobilize inner resources and strength of the student just before entering the examination circuit.
  Other Names: Resources and inner strength mobilization
  Arms: Inner resource mobilization
Other: Control — 6 minutes of standardized neutral video on general topics that generates no modification of affects just before entering the examination circuit.
  Other Names: Standardized video
  Arms: Control

SUMMARY:
Objective Structured Clinical Examination (OSCE) is a newly implemented evaluation standard for medical students and is a determinant part of the national competition they have to undergo.

Exam periods are significantly associated with increased stress and anxiety which led to reduced performance, impaired memorization and impaired workload capacities.

Cardiac biofeedback and mindfulness techniques are efficient methods for stress reduction. Interventions that aim to mobilize competence, such as mobilization of inner strength and resources techniques, should improve the level of preparation of medical students. These three procedures could influence the stress level and improve performance during the OSCE.

There is currently no study exploring the effect of these physiological and psychological procedures on the performance during OSCE for medical students.

DETAILED DESCRIPTION:
This randomized, controlled, monocentric study will take place during mandatory rehearsal of Objective Structured Clinical Examination for third year medical students. For examination purposes, the students will be divided into four groups that will undergo identical exams at the same time in four parallel circuits.

Before entering the station of OSCE and before being involved in the research, all the students will receive information about the study and sign a consent form.

Participants will undergo short questionnaires regarding inner resources available to accomplish the exam and questionnaire exploring self-confidence.

Then the groups of students will be randomized in four intervention groups before the examination circuit. All the interventions will last six minutes long. The randomization groups are:

* Cardiac biofeedback (guided through a video with a breathing cursus and visual cardiac feedback)
* Mindfulness (guided through a video)
* Resources and Inner Strength Mobilization (guided through a video)
* Control group (guided through a neutral-content video)

At the end of the intervention, all the students will undergo short questionnaires regarding their perceived level of resources to accomplish the exam and their self-confidence.

During the OSCE, examiner will evaluate the performance of the students. All the examiner will be blind to the student's experimental group.

After the OSCE circuit, students will be asked to rate their perceived emotional performance during the exam (Likert scale). They have to answer a visual analogue scale, to declare how they estimate that the intervention has influenced their performance (from negative to positive).

The final score of the student, as determined by the examiner, will be composed of:

* Objective quantitative score with respect to the specific evaluation grid for each OSCE scenario.
* Subjective qualitative score (Likert scale)

Emotional Performance will be assessed by two means:

* Emotional performance score hetero-evaluated by the examiner (Likert scale)
* Emotional performance score auto-evaluated by the student (Likert scale) Main objective is to show that a preventive physiological and psychological intervention (cardiac biofeedback, or mindfulness, or Inner resource mobilization) is better than a neutral-content video on the following performance during OSCE.

The main outcome is the mean score of student objective quantitative score (composed by the mean of each quantitative score of the five stations during the OSCE) at as determined by the university examiner.

Secondary objectives are to compare the effects of the interventions on all the components of the performance score: objective quantitative score, subjective qualitative score, emotional performance score hetero and auto-evaluated. Three sub-scores of the objective quantitative score (divided into communication (C), knowledge (K) and Skills (S) performance) will be compared. Visual analogue scales of perceived inner resource available to pass the exam, self-confidence and perceived effect of the intervention on the performance will also be compared.

ELIGIBILITY:
Inclusion Criteria:

* Adult person
* Registered as medical student at the university
* Participating at OSCE examination
* Have signed an informed consent form.

Exclusion Criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 490 (Actual)
Dates: Start 2022-05-17 (Actual); Primary Completion 2022-07-19 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Mean of quantitative performance score for all the exam | rated during the exam, calculated during the first 2 weeks after the exam
  Mean of quantitative performance score for all the exam (mean of the five performance score for the 5 stations of the exam (from zero to maximum: 40). Each objective performance score of a station is determined by a specific scenario grid performance.) The primary outcome will be determined by university examiners who are independent of the study and blinded to the interventions.

SECONDARY OUTCOMES:
Mean Differences in Subjective Performance | rated during the OSCE, calculated during the first 2 weeks after the OSCE
  The subjective qualitative performance is the score qualitative of overall performance of each student as determined by university examiners who are independent of the study and blind to the intervention (mean of 5 scores). Each score of subjective performance will be determine on a Likert scale (from 0 to 5).
Mean Differences in Three Objective Performance sub-scores | rated during the exam, calculated during the first 2 weeks after the exam
  Each scenario has a specific grid composed of numerous items. Each item of all the scenario grid will be sorted by regarding if they evaluate communication ability (C), knowledge (K), or skills ability (S).
  The sorting of the items between the three groups (C, K and S) will be assessed by two experts independently. In case of a disagreement, a third expert will be asked to choose. Every student will get a score regarding these three sub-scores (from 0 to maximum: 40)
Mean Differences in Hetero-Evaluated Emotional Performance | Once - in the 2 minutes after the OSCE station
  The emotional performance rated by examiners is the overall appreciation of the student ability to control his/her emotion during each station (e.g., control stress, communicate with empathy…). For each OSCE station, the student emotional performance will be evaluated on a Likert scale (0 to 5) by the examiner.
Mean Differences in Auto-evaluated Emotional Performance | during the first 5 minutes just after OSCE
  The emotional performance rated by the student himself is the overall appreciation of the student demonstrated ability during the whole OSCE (the five stations) to control his/her emotion (e.g., control stress, communicate with empathy…). Each student will evaluated his/her performance on a Likert scale (0 to 5).
Mean Difference of Inner Resource | Two times : 10min before OSCE (before intervention) and just 2 minutes before the OSCE (after intervention)
  Numerical VAS on inner resource available perceived (from 0 to 100 : maximum)
Mean difference of perceived impact of the intervention on performance | Just 5 minutes after the OSCE
  Numerical Visual analog scales (VAS) on perceived impact of the intervention on performance (from zero: negative to 100: positive)
Mean Differences of Self confidence | Two times : 10min before OSCE (before intervention) and just 2 minutes before the OSCE (after intervention)
  Numerical VAS on self-confidence perceived from zero to 100: maximum

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Rode, Ph. D., Study Chair — Claude Bernard University; Marc Lilot, Ph. D., Study Director — Claude Bernard University
Locations (1):
- Claude Bernard University, Lyon, France

REFERENCES:
- [Derived] Schlatter S, Berland A, Lutz A, Shankland R, Barret N, Guillaumee T, Duclos A, Cortet M, Rimmele T, Rode G, Lilot M. Effect of coping interventions on performance of medical students during objective structured clinical examination: A randomized controlled trial. Med Teach. 2025 Aug;47(8):1367-1376. doi: 10.1080/0142159X.2024.2431137. Epub 2025 Jan 3. PMID 39752249